CLINICAL TRIAL: NCT03568136
Title: A Randomized, Placebo-controlled, Double-blind Study to Scrutinize the Efficacy of Secukinumab in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Investigation of Efficacy of Secukinumab in Patients With Moderate to Serve Atopic Dermatitis
Acronym: Secu_in_AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Secu_Trial; 2016-005181-57 (EudraCT Number)
Record Dates: First submitted 2018-05-23; First posted 2018-06-26 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2020-05

CONDITIONS: Dermatitis, Atopic; Eczema, Atopic; Neurodermatitis, Atopic
Keywords: neurodermatitis; moderate to severe inflammatory reaction of the skin; Skin and Connective Tissue Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Neurodermatitis; Skin and Connective Tissue Diseases | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Experimental): Patients in treatment arm A receive 300 mg Secukinumab administered as 2 subcutaneous injections of 150 mg (i.e. 2x 150 mg) at baseline day 1 and week 1, 2, 3, 4, 8, 12 and injections with placebo at week 5, 6, 7 and 16. For assessments of the study endpoints were followed up visits at week 20 and 24. Placebo will be administered as 2 subcutaneous injections.
  Interventions: Drug: Secukinumab 300 mg; Drug: Placebo
- Treatment Arm B (Placebo Comparator): Patients in treatment arm B receive placebo until visit 3 (week 3) and will switch to Secukinumab 300 mg s.c. up from visit 4 (week 4), visit 5, 6, 7, 8, 12 and16. For assessments of the study endpoints were followed up visits at week 20 and 24.
  Interventions: Drug: Secukinumab 300 mg; Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab 300 mg — Solution for injection in pre-filled syringe
  Other Names: COSENTYX ®
Drug: Placebo — Solution for injection in pre-filled syringe
  Other Names: Placebo (for Secukinumab)

SUMMARY:
The overall aim of this study is to assess the effects of a new treatment called Secukinumab in adults suffering from moderate to severe atopic dermatitis. Furthermore, the study shall support the extension of the approval for Secukinumab from psoriasis to atopic dermatitis. The effectiveness of Secukinumab is determined on the reduction of the eczema score EASI 50 (Eczema Area and Severity Index, a tool to measure the severity of atopic dermatitis) at week 4.

DETAILED DESCRIPTION:
Secukinumab is a humanized anti-IL-17A monoclonal antibody. Since Secukinumab is well established in the therapy of psoriasis with a highly favorable benefit to risk ration and IL-17 has been described in atopic dermatitis this study aims to investigate the effects of anti-IL-17 in atopic dermatitis.

This is a randomized, placebo-controlled, multicenter, double-blinded study to evaluate the efficacy and safety of subcutaneous Secukinumab compared to placebo in 45 adults with atopic dermatitis.

The study consists of 3 periods: a screening period of at least -14 days and up to -35 days, and a treatment period of 16 weeks and a follow-up period of additional 8 weeks. During the screening period eligibility of the patients is confirmed. Eligible patients are randomized 2:1 to treatment arm A or B at Day -7 (+2 to -15) during the randomization visit. Secukinumab (Cosentyx®) will be used according to the official label and SmPC (Summary of Product Characteristics). Patients in treatment arm A receive 300 mg Secukinumab administered as 2 subcutaneous injections of 150 mg (i.e. 2x 150 mg) at baseline day 1 and week 1, 2, 3, 4, 8, 12 and injections with placebo at week 5, 6, 7 and 16. For assessments of the study endpoints visits are performed at weeks 20 and 24. Placebo will be administered as 2 subcutaneous injections. Patients in treatment arm B receive placebo until visit 3 (week 3) and will switch to Secukinumab 300 mg s.c. up from visit 4 (week 4), visit 5, 6, 7, 8, 12 and16. For assessments of the study endpoints visits are performed at weeks 20 and 24.

ELIGIBILITY:
Inclusion Criteria:

1. Atopic dermatitis (intrinsic disease without IgE mediated sensitization defined by negative history and negative SX-1 CAP FEIA or extrinsic disease defined by positive history and / or positive SX-1 CAP FEIA),
2. SCORAD index score ≥ 25,
3. EASI ≥ 16,
4. Male and female patients at the age of 18 to 85 years,
5. Signed Informed Consent,
6. Subjects must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study related activity is performed,
7. Subject is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, and physical examination,
8. Patients with stable chronic asthma, treated with inhaled corticosteroids, will be allowed to participate.

Exclusion Criteria:

1. Other inflammatory skin disease than atopic dermatitis,
2. Use of cyclosporine, azathioprine, mycophenolate [wash-out period of 4 weeks]; Phototherapy (PUVA, NB-UVB, UVA1; [wash-out period of 2 weeks]), Dupilumab (Dupixent®; [wash-out period of 12 weeks])
3. Subjects expected to be exposed to an undue safety risk if participating in the trial including chronic infections,
4. Contraindications of Secukinumab by label (i.e. approval for the treatment of psoriasis in the EU - refer to point 14 - 16 at the bottom of this section),
5. Current severe progressive or uncontrolled disease which in the judgment of the investigator renders the subject unsuitable for the trial,
6. Plans for administration of live vaccines during the study period,
7. Chronic infection,
8. Patients with instable chronic asthma,
9. Any chronic inflammatory bowel disease (e.g. Crohn's disease),
10. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>10 mIU/mL),
11. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unwilling to use effective contraception during the study and for 20 weeks after stopping treatment. Effective contraception is defined as either:

    1. Barrier method: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicide (where available). Spermicides alone are not a barrier method of contraception and should not be used alone,

       The following methods are considered more effective than the barrier method and are also acceptable:
    2. Total abstinence: When this is in line with the preferred and usual lifestyle of the subject (Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception),
    3. Female sterilization: have had a surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment,
    4. Male partner sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject,
    5. Use of established oral, injected or implanted hormonal methods of contraception, intrauterine device (IUD) or intrauterine system (IUS) NOTE: Women are considered post-menopausal and not of child bearing potential if they have had:

    i. 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or • six months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL

    Or

    ii. Surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
12. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening,
13. Positive with hepatitis B surface antigen (HBsAg) or hepatitis C antibody at the screening visit (a report ≤ 6 months is also accepted),
14. History of alcohol or drug abuse within 1 year of the screening visit,
15. Planned major surgical procedure during the patient's participation in this study,
16. Hypersensitivity against Secukinumab,
17. Active or reactive tuberculosis,
18. Participation in other clinical studies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Reduction in EASI | week 4 (visit 4)
  Proportion of patients with a reduction of the eczema score EASI of at least 50%. The proportions are then compared between study arms.

SECONDARY OUTCOMES:
Reduction of EASI | baseline (day 1, visit 0) and End of Trial (Arm A week 12 / Arm B week 16)
  To compare the proportions of patients with a reduction of the eczema score EASI 50.
Reduction of EASI | Arm A week 12 / Arm B week 16
  To compare the number of patients with a reduction of the eczema score EASI 50.
Reduction in SCORAD (Scoring atopic dermatitis) | day 1, week 4 and Arm A week 12 / Arm B week 16
  The number of patients with a reduction of 50 % in SCORAD index.
Change in pruritus score (Visual Analogue Scale) | day 1, week 4 and Arm A week 12 / Arm B week 16
  To compare the proportion of patients with change in pruritus score (VAS) by 50 %.
Change in IGA Score (5-point Investigator's Global Assessment) | Arm A week 12 / Arm B week 16
  To compare the proportion of patients who achieve a score of "clear-0" or "almost clear-1" in the static IGA score compared to baseline.
Serum biomarkers CCL17 and CCL22 | day 1, week 4 and Arm A week 12 / Arm B week 16
  To compare the serum biomarkers CCL17 and CCL22.
Increase in DLQI (Dermatology Life Quality Index) | day 1, week 4 and Arm A week 12 / Arm B week 16
  To compare the proportion of patients achieving increase in DLQI by 30 %.
Consumption of topical methylprednisolone aceponate | day 1, week 4 and Arm A week 12 / Arm B week 16
  To evaluate the quantification of the consumption of topical methylprednisolone aceponate 0.1% in gram.
Serious and non-serious adverse drug reactions | treatment phase (day 1 up to week 16), follow-up phase (week 20, week 24)
  To observe any serious adverse drug reactions and non-serious adverse drug reactions.
Gender distribution in patients with atopic dermatitis | study arm A week 4 and both study arms week 16
  Subgroup analyses will be performed to compare the effects of treatment with Secukinumab in male and female patients. Therefore, the recorded gender data will be used and separately analyzed for the above mentioned primary and secondary endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Beissert, Prof. Dr., Principal Investigator
Locations (5):
- Germany (5):
  - Klinische Forschung Dresden GmbH, Dresden
  - Carl Gustav Carus University Hospital, Department of Dermatology, Dresden
  - SRH Wald-Klinikum Gera, Center for Clinical Studies, Gera
  - Hannover Medical School, Department for Dermatology, Allergy and Venereology, Hanover
  - SIBAmed Studienzentrum GmbH & Co KG, Leipzig

IPD SHARING:
Plan to Share IPD: No